CLINICAL TRIAL: NCT02029937
Title: High Resolution Microendoscopy for the Detection of Esophageal Squamous Cell Neoplasia: A Randomized, Multicenter Trial of Accuracy, Yield, and Clinical Impact
Brief Title: High Resolution Microendoscopy for the Detection of Esophageal Squamous Cell Neoplasia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anandasabapathy, Sharmila, M.D. (Individual)
Collaborators: William Marsh Rice University (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GCO 13-0396
Record Dates: First submitted 2013-12-17; First posted 2014-01-08 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Suspected or Known Squamous Cell Neoplasia; Prior History of Squamous Cell Dysplasia and /or Neoplasia
Keywords: Squamous cell neoplasia; Proflavine; Lugol's chromoendoscopy
MeSH Terms: conditions — Neoplasms | interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proflavine, high resolution imaging (Experimental): 5-10 ml of proflavine hemisulfate (0.01%) will be sprayed on the esophageal mucosa. The HRME will then be inserted through the endoscope and gently placed against the mucosa. Imaging of abnormal tissues will be performed.
  Interventions: Drug: Proflavine, high resolution imaging
- Standard of care (No Intervention): No invention

INTERVENTIONS:
Drug: Proflavine, high resolution imaging — 5-10 ml of proflavine hemisulfate (0.01%) will be sprayed on the esophageal mucosa. The HRME will then be inserted through the endoscope and gently placed against the mucosa. Imaging of abnormal tissues will be performed.
  Other Names: Proflavine hemisulfate
  Arms: Proflavine, high resolution imaging

SUMMARY:
The overall objective of this multicenter trial is to determine whether the use of a low-cost, high-resolution microendoscope during diagnostic upper endoscopy can improve the efficiency and accuracy of endoscopic screening for esophageal squamous cell neoplasia. This is a multicenter clinical trial of a novel technology, a miniaturized, lower cost (< $3, 500) microscope device which can be used during upper endoscopy to image the gastrointestinal epithelium. This high-resolution microendoscope (HRME) was developed by our collaborators at RICE University and provides >1000X magnified images of the esophageal mucosa.

DETAILED DESCRIPTION:
Our central hypothesis is that HRME can improve the efficiency and clinical impact of endoscopic screening and surveillance of esophageal squamous cell neoplasia by providing in-vivo optical biopsies comparable to standard histology. Specifically, HRME will allow more detailed evaluation of Lugol's abnormal areas, allowing selective biopsy or removal of neoplastic mucosa. We hypothesize that this will improve the accuracy and diagnostic yield of mucosal sampling.

We also hypothesize the HRME will provide additional, more accurate information regarding the presence of neoplasia that will impact upon the physician's decision to obtain a mucosal biopsy or perform endoscopic therapy (endoscopic mucosal resection or ablation). This could potentially minimize the number of unnecessary biopsies and enable the physician to perform endoscopic therapy at the time of the initial examination, rather than delaying endoscopic treatment to another procedure following pathologic confirmation of the initial biopsies.

Primary Aims:

1. To compare the efficiency of HRME + Lugol's chromoendoscopy (HRME + LC) to that of Lugol's chromoendoscopy alone (LC) for the diagnosis of esophageal squamous cell neoplasia. Efficiency will be defined as:

   1. Diagnostic Yield: The number of neoplastic biopsies/total number of biopsies obtained in patients who receive biopsies.
   2. 'Patients saved': # patients who receive no biopsies
   3. Procedure time: Total procedure time in the HRME-LC arm compared to the LC arm.
2. To prospectively determine the potential clinical impact of HRME + Lugol's chromoendoscopy (HRME-LC) to Lugol's Chromoendoscopy (LC) by determining if HRME changes the decision to perform endoscopic therapy (endoscopic mucosal resection or ablation) or perform a mucosal biopsy.
3. To prospectively compare the performance characteristics of HRME-LC to LC for the prediction of squamous esophageal neoplasia in flat mucosa and mucosal lesions using histopathology as the gold standard:

   (a) To determine the sensitivity, specificity, positive and negative predictive value for the identification of neoplasia on a per biopsy and per patient analysis
4. To determine the cost-effectiveness of HRME-LC to LC alone for the endoscopic screening and surveillance of esophageal squamous neoplasia in the US and China.

ELIGIBILITY:
Inclusion Criteria:

All inclusive outpatients undergoing routine (standard of care) Lugol's chromoendoscopic evaluation for suspected or known squamous cell neoplasia will be enrolled as well as any outgoing patients referred to the clinic with any prior history of squamous cell dysplasia and/or neoplasia will also be considered eligible as they will serve as study population for the surveillance group.

Exclusion Criteria:

* Allergy or prior reaction to the fluorescent contrast agent proflavine
* Patients who are unable to give informed consent
* Known advanced squamous cell carcinoma of the distal esophagus, or dyplastic/suspected malignant esophageal lesion greater than or equal to 2cm in size not amenable to endoscopic therapy
* Patient unable to undergo routine endoscopy with biopsy:
* women who are pregnant or breastfeeding
* prothrombin time greater than 50% of control; PTT greater than 50 sec, or INR greater than 2.0
* inability to tolerate sedated upper endoscopy due to cardio-pulmonary instability or other significant medical issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the efficiency of HRME+Lugol's chromoendoscopy (HRME+LC) to that of Lugol's chromoendoscopy alone (LC) for the diagnosis of esophageal squamous cell neoplasia. | 1 day
  Efficiency
  1. Diagnostic yield: The number of neoplastic biopsies/total number of biopsies obtained in patients who received biopsies.
  2. 'Patient saved': # of patients who received no biopsies
  3. Procedure time: Total procedure time in the HRME-LC arm compared to the LC arm.

SECONDARY OUTCOMES:
Determination whether HRME changes the decision to perform endoscopic therapy or perform a mucosal biopsy | 1 day
  Clinical Impact

OTHER OUTCOMES:
Comparison of the performance characteristics of HRME to LC for the prediction of squamous esophageal neoplasia using histopatholgy as the gold standard. The cost-effectiveness of HRME-LC to LC alone. | 1 day
  Cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Anandasabapathy, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- Baylor College of Medicine, Houston, Texas, United States
- China (2):
  - First Hospital of Jilin University, Changchun, Jilin
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences (CICAMS), Beijing

REFERENCES:
- [Derived] Tan MC, Li Z, Patel KK, Zhang F, Yu X, Wang X, Rosen DG, Dawsey SM, Xue L, Hur C, Schwarz RA, Vohra I, Tang Y, Wu M, Wang T, Carns J, Xu H, Richards-Kortum RR, Wang G, Anandasabapathy S. A High-Resolution Microendoscope Improves Esophageal Cancer Screening and Surveillance: Implications for Underserved Global Settings Based on an International Randomized Controlled Trial. Gastroenterology. 2025 Mar;168(3):496-507.e3. doi: 10.1053/j.gastro.2024.10.025. Epub 2024 Oct 29. PMID 39477026

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT02029937/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT02029937/ICF_001.pdf